CLINICAL TRIAL: NCT05592405
Title: Nociplastic Pain Measurement and Sensory Profiles in Patients with Acute and Chronic Low Back Pain: a Longitudinal Observational Cohort Study
Brief Title: Nociplastic Pain Symptoms and Sensory Profiles in Low Back Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Pieter Graper, Principal investigator, Vrije Universiteit Brussel
Other Study IDs: QST_SPs
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Central Sensitisation; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Assessing associations between Sensory profiles and nociplastic pain symptoms, and assessing the prognostic value of sensory profiles in the development of nociplastic pain symptoms in a low back pain population.

DETAILED DESCRIPTION:
Therefore, the investigators aims are:

* The primary aim of the study is to assess associations between Sensory Profiles (Adolescent/Adult Sensory Profiles) and Nociplastic pain Symptoms, in the acute and chronic low back pain population.
* The secondary aim is to assess the prognostic value of sensory profiles in the transition to central sensitisation and pain, in the acute and chronic low back pain population at twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-specific LBP
* with or without radiating pain
* aged 18-65 years
* able to read and understand the Dutch language

Exclusion Criteria:

* previous lumbar spinal surgery
* radiculopathy or any specific cause of low back pain such as lumbar spinal stenosis, current malignancy, spondyloarthropathy, osteoporosis, spondylolisthesis, major trauma, infection, or systemic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Evaluation of eligibility will take place during assessment when the participant reports in primary care physiotherapy practice for the treatment of LBP.
  Patients will be included consecutively and measurements will be obtained by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Central sensitiszation QST | 12 weeks follow-up
  Quantitative sensory testing
Central senzitization CSI | 12 weeks follow-up
  Central sensitization inventory
Central sensitization PSQ | 12 weeks follow-up
  Pain sensitization questionnaire

OTHER OUTCOMES:
Demograpics | 12 weeks
  established prognostic factors for low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Scafoglieri, PhD, Study Director — Vrije Universiteit Brussel
Locations (1):
- Fysiomobilae, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Sharing is unlikely as the data set includes pseudo-anominizised highly confidential data, of which the participants do not gave their consent to use their provided data.